CLINICAL TRIAL: NCT06283056
Title: Radiofrequency Microneedling With Multi-Depth Targeting Per Insertion for The Treatment of Cellulite
Brief Title: RF Microneedling With Multi-Depth Targeting Per Insertion for The Treatment of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO611073A
Record Dates: First submitted 2023-11-16; First posted 2024-02-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: Cellulitis of Leg

STUDY DESIGN:
Intervention Model Description: Prospective, open-label clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Treatment (Experimental): Eligible subjects will undergo two treatments with the Morpheus8 device using the 3, 5 7 mm depths or sequential (Burst) mode, based on the treating physician's discretion.
  Interventions: Device: Device treatment

INTERVENTIONS:
Device: Device treatment — InMode RF system with Morpheus8 Body (up to 7mm depth) Eligible subjects will undergo two treatments with the Morpheus8 device using the 3, 5 7 mm depths or sequential (Burst) mode, based on the treating physician's discretion..each subject is approximately 9 months (including screening, two treatments (2 months apart) and 3 follow-up visits at 1 month, 3 months, and 6 months post treatment.

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of Morpheus 8 Body 40-pin tip up to 7mm depth Applicator for subdermal treatment of cellulite appearance, skin laxity, and subcutaneous fat deposits.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the safety and efficacy of Morpheus 8 Body 40-pin tip up to 7mm depth Applicator for subdermal treatment of cellulite appearance, skin laxity, and subcutaneous fat deposits.

Prospective, open-label, baseline-controlled, clinical study to evaluate the Morpheus8 device for treatment of cellulite, skin laxity, and subcutaneous fat deposits of the thighs.

Eligible subjects will undergo two treatments with the Morpheus8 device using the 3, 5 7 mm depths or sequential (Burst) mode, based on the treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18-65 (inclusive)
* BMI interval: 18.5 ≤ BMI ≤ 30 (normal to overweight, but not obese).
* Subject having cellulite grade 1-4 as graded using the Clinician Reported Photonumeric Cellulite Severity Scale (CR-PCSS)7.
* The patients should understand the information provided about the treatment, possible benefits and side effects, and sign the Informed Consent Form, (including the permission to use photography).
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods (i.e liposuction, any cellulite/circumference reduction treatments using medical devices, etc.) in the treatment area for the last 6 months and during the entire study period.
* Females of Childbearing potential must be using an approved method of birth control. Subjects who are capable of becoming pregnant will undergo a urine pregnancy test.

Exclusion Criteria:

* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Superficial permanent implant in the treated area such as metal plates and screws, metal piercing, silicone implants or an injected chemical substance.
* Known sensitivity/allergy to Lidocaine
* Current or history of skin cancer (remission of 5 years), or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing or lactating.
* History of bleeding coagulopathies or use of anticoagulants.
* Chronic or current use of NSAIDs or other anti-inflammatory therapies (e.g., Ibuprofen, etc.)
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Any uncontrolled medical condition (i.e., endocrine disorders, diabetes, thyroid disfunction or hormonal virilization) that in the opinion of the investigator, the subject's safety may be compromised.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Any surgery or treatment such as laser or chemicals in treated area within 3-6 months prior to treatment or before complete healing.
* Any medical condition that in the opinion of the investigator, such condition would compromise the safety of the subject or quality of the study data.
* Current, or past participation in a clinical trial within the past 30 days.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 40 female subjects aged 18-65 seeking cellulite treatment. Treatment areas include: thighs.
Enrollment: 48 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Cellulite assessment based on Clinician Reported Photonumeric Cellulite Severity Scale | 6 Months
  Cellulite assessment based on Clinician Reported Photonumeric Cellulite Severity Scale (using pre (baseline) and post treatment Standard medical photography, having at least mean of one-unit improvement (1-point score reduction).
  0 - None - No evident cellulite
  1. - Almost none - A few superficial dimples or ridges
  2. - Mild - Several dimples or ridges, of which most are superficial
  3. - Moderate - Many dimples or ridges, of which more are somewhat deep
  4. - Severe - A lot of dimples or ridges, of which many are deep, covering most of the skin area
Cellulite assessment based on DiBernardo Photonumeric Cellulite Severity Scale | 6 Months
  Cellulite assessment based on DiBernardo Photonumeric Cellulite Severity Scale using pre (baseline) and post-treatment Standard medical photography, having at least a mean of one-unit improvement (1-point score reduction).
  This 5-point photo numeric scale rates cellulite severity from "0" (none) to "4" (severe) from a clinician's perspective

SECONDARY OUTCOMES:
Subject assessment of improvement | 1 month
  Subject assessment of improvement using 0 - 4 -points Likert scale at 1 month, 3 months, 6 months follow up visits:
  4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No change
Subject assessment of improvement | 3 months
  Subject assessment of improvement using 0 - 4 -points Likert scale at 1 month, 3 months, 6 months follow up visits:
  4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No change
Subject assessment of improvement | 6 months
  Subject assessment of improvement using 0 - 4 -points Likert scale at 1 month, 3 months, 6 months follow up visits:
  4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No change
Subject assessment of satisfaction | 1 month
  Subject assessment of satisfaction will be filled-out by subjects only using 4-points Likert scale at 1 month, 3 months, 6 months follow up visits:
  +2 = Very satisfied; +1 = Satisfied; -1 = Dissatisfied; -2 = Very Dissatisfied
Subject assessment of satisfaction | 3 months
  Subject assessment of satisfaction will be filled-out by subjects only using 4-points Likert scale at 1 month, 3 months, 6 months follow up visits:
  +2 = Very satisfied; +1 = Satisfied; -1 = Dissatisfied; -2 = Very Dissatisfied
Subject assessment of satisfaction | 6 months
  Subject assessment of satisfaction will be filled-out by subjects only using 4-points Likert scale at 1 month, 3 months, 6 months follow up visits:
  +2 = Very satisfied; +1 = Satisfied; -1 = Dissatisfied; -2 = Very Dissatisfied
Investigator assessment of the skin appearance improvemen | 1 month
  Investigator assessment of the skin appearance improvement comparing pre and post treatment using Global aesthetic improvement 4-point grading scale (0=No tightening/firmness, 1= Slightly visible tightening/firmness, 2= Visible tightening/firmness, 3= Very visible tightening/firmness) at all follow up visits.
Investigator assessment of the skin appearance improvement | 3 months
  Investigator assessment of the skin appearance improvement comparing pre and post treatment using 0 - 4 -points Likert scale at 1 month, 3 months, 6 months follow up visits:
  4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No difference
Investigator assessment of the skin appearance | 6 months
  Investigator assessment of the skin appearance improvement comparing pre and post treatment using 0 - 4 -points Likert scale at 1 month, 3 months, 6 months follow up visits:
  4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No difference
Investigator assessment of the cellulite following subdermal Morpheus8 treatment | 1 Month
  Statistically significant improvement in global aesthetic appearance of cellulite, as assessed by PI using Global aesthetic improvement 5-point grading scale (0=No change, 1=1%-24%%, 2=25%-49%, 3=50%-74% improvement, and 4=75%-100%)
Investigator assessment of the cellulite following subdermal Morpheus8 treatment | 3 Months
  Statistically significant improvement in global aesthetic appearance of cellulite, as assessed by PI using Global aesthetic improvement 5-point grading scale (0=No change, 1=1%-24%%, 2=25%-49%, 3=50%-74% improvement, and 4=75%-100%)
Investigator assessment of the cellulite following subdermal Morpheus8 treatment | 6 Months
  Statistically significant improvement in global aesthetic appearance of cellulite, as assessed by PI using Global aesthetic improvement 5-point grading scale (0=No change, 1=1%-24%%, 2=25%-49%, 3=50%-74% improvement, and 4=75%-100%)

OTHER OUTCOMES:
Adverse Event rate | For the duration of the study
  Rate of all device and procedure related adverse events (AE's) and serious adverse events (SAE's) occurring during the study
Pain Scale | Immediately post each procedure
  Pain assessment will be performed immediately post treatment using Numeric Pain Rating Scale (NPRS) from 0 to 10. 0 = no pain 10 - worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: . Macrene Alexiades, md, Principal Investigator; Rod Rohrich, md, Principal Investigator
Locations (2):
- United States (2):
  - Dermatology & Laser Surgery Center of New York, New York, New York
  - Dallas Plastic Surgeon, Dallas, Texas